CLINICAL TRIAL: NCT00651885
Title: A Randomized, Single-Center, Placebo Controlled Study To Assess the Safety of UT-15C (Treprostinil Diethanolamine) Sustained Release (SR) in Patients Undergoing an Infra-Popliteal Endovascular Intervention for the Treatment of Critical Limb Ischemia
Brief Title: Safety Study of UT-15C SR (Oral Treprostinil) in Patients Undergoing a Lower Limb Endovascular Procedure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2006.219.B
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Critical Limb Ischemia
Keywords: UT-15C; Peripheral Vascular Disease; Treprostinil
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Vascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 arm (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 arm (Experimental): treprostinil dienthalomine
  Interventions: Drug: treprostinil dienthanolmine sustained release

INTERVENTIONS:
Drug: treprostinil dienthanolmine sustained release — UT-15C SR 1mg tablet
  Other Names: UT-15C SR
  Arms: 1 arm
Drug: Placebo — Placebo
  Arms: 2 arm

SUMMARY:
In chronic CLI patients who are appropriate candidates for endovascular procedures - and many patients are not because of their advanced age and disease state - the treatment regimen may include endovascular procedures such as percutaneous transluminal endovascular intervention, as well as reconstructive surgical procedures such as grafts or bypasses. Amputation is a last resort where limb salvage cannot be achieved. Despite the success of percutaneous intervention for small coronary vessels with lumen diameters less than 3 mm, similar techniques have had limited success in the lower extremity vessels. Infra-popliteal, or below the knee endovascular intervention, is commonly plagued by subacute thrombotic closure and restenosis in as many as 50% of treated patients. As a result of the limited success, these percutaneous procedures have been reserved for the severest cases whereby limb loss is imminent without intervention. In this context, the sickest of all patients are enrolled in these trials and poor outcomes are common regardless of the intervention. Agents that promote intracellular cAMP accumulation, including prostacyclin analogues and phosphodiesterase inhibitors, suppress smooth muscle proliferation, promote vasodilatation and inhibit platelet aggregation. These properties suggest that prostacyclin analogues such as treprostinil will be useful adjuncts to peripheral endovascular intervention and perhaps increase the number of patients with CLI that can benefit from peripheral endovascular intervention. An orally available prostacyclin analogue could represent an important treatment advance in the prevention of restenosis following infrapopliteal angioplasty. In the present study, the safety and efficacy of oral UT-15C sustained release (SR) tablets will be compared to placebo in patients with CLI undergoing an infra-popliteal endovascular intervention.

DETAILED DESCRIPTION:
This study is a randomized, placebo controlled, single-center, evaluation of the safety and efficacy of UT-15C SR compared to placebo in patients with CLI with a planned infra-popliteal endovascular intervention procedure. Conventional therapy should be continued for all patients in the study. Conventional therapy is defined as the customary best medical practice at this investigative site for CLI, including analgesics for rest pain, debridement and wound care for ischemic wounds, etc., as long as such care meets the other requirements of the study and does not include prohibited therapies or investigational medications. A total of 20 patients will be prospectively randomized (1:1) to conventional treatment and placebo therapy in conjunction with an endovascular procedure or conventional treatment and UT-15C SR therapy in conjunction with an infrapopliteal endovascular procedure. Treatment is UT-15C sustained release (SR) tablets (1.0 mg dosage strength) or placebo. Treatment will be initiated at 1 mg twice daily with dose escalation of an additional 1 mg twice daily every 5 days if clinically indicated based upon the presence of known prostacyclin adverse events or adverse events that in the opinion of the investigator are attributable to UT-15C SR. Doses should be maximized throughout the Treatment Phase up to a maximum dose of 5 mg twice daily at the end of 12-weeks. Patients will return to the institution for the endovascular procedure at least 4 days after starting study drug and continue study drug, throughout the endovascular procedure and to Week 12. All patients will return to the clinic at Weeks 2, 6 and 12 for Treatment Phase assessments, and then Weeks 26 and 52 for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 or older.
2. Have an anticipated infra-popliteal endovascular intervention.
3. Have a diagnosis of stage IIb- IVa (Fontaine) or stage 3- 5 (Rutherford scale) CLI due to documented peripheral arterial disease (Appendix E)
4. If female, be physiologically incapable of childbearing or practicing acceptable methods of birth control.
5. Have signed an appropriate informed consent for participation in this study.

Exclusion Criteria:

1. Have had a previous endovascular intervention or stenting on the target limb.
2. Be hemodynamically unstable, on hemodialysis for end stage renal failure, or have acute renal, cardiac or pulmonary failure.
3. Have a history of intracranial bleeding, bleeding ulcer, urinary tract bleeding; or bleeding due to significant trauma within six weeks prior to study entry.
4. Have a life-threatening malignancy requiring aggressive chemotherapy.
5. Have any condition or laboratory value which, based on information in the UT-15C SR investigators' brochure, would constitute an unacceptable risk to the patient's safety, in the opinion of the investigator.
6. Have unstable psychiatric status or be mentally incapable of understanding the objectives, nature or consequences of the trial.
7. Have a known hypersensitivity to prostacyclin.
8. Have participated in any investigational trial within 30 days of study drug initiation.
9. Have been a non-responder to chronic (>30 days) prostanoid treatment, or have completed a chronic trial of prostanoid therapy within 30 days of study drug initiation.
10. Be a pregnant or nursing woman.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess the tolerability and safety of UT-15C SR as compared to placebo tablets in subjects with critical limb ischemia (CLI) undergoing an infra-popliteal endovascular intervention procedure. | 12 weeks

SECONDARY OUTCOMES:
To assess the efficacy of UT-15C SR as compared to placebo tablets on measures of clinical outcomes in subjects with critical limb ischemia (CLI) undergoing an infra-popliteal endovascular intervention procedure. | 12-52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Grise, M.D., Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States